CLINICAL TRIAL: NCT06953791
Title: Comparison of Quality of Life During a Flare of Crohn's Disease Treated With Standard of Care or an Adapted Crohn's Disease Exclusion Diet With Partial Enteral Nutrition in Adult Patients
Brief Title: Comparison of Quality of Life During a Flare of Crohn's Disease Treated With Prednisolone or aCDED With PEN in Adult Patients
Acronym: CONSISTENT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONSISTENT
Record Dates: First submitted 2024-01-04; First posted 2025-05-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease; Nutrition Assessment; Diet Therapy
Keywords: Nutrition; crohn disease; diet therapy; consistent
MeSH Terms: conditions — Crohn Disease | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Prednisolone
  Interventions: Drug: Prednisolone
- Interventional arm (Experimental): Adapted Crohn's disease Exclusion Diet (aCDED)
  Interventions: Dietary Supplement: aCDED + Modulen

INTERVENTIONS:
Dietary Supplement: aCDED + Modulen — Unique diet + partial enteral nutrition (PEN): This group will receive as follows:
  * Weeks 1-6: 50% of dietary needs from PEN (Modulen, ModuLife phase I) and 50% from a limited whole food diet
  * Weeks 7-12: 25% of dietary needs from PEN (Modulen, ModuLife phase II) and 75% from a limited whole food diet
  * Weeks 12-48: liberal diet and Modulen as needed
  Arms: Interventional arm
Drug: Prednisolone — 1 mg/kg, tapering scheme
  Arms: Standard of care

SUMMARY:
Crohn's disease (CD), a type of inflammatory bowel disease (IBD), is on the rise globally. Although medical treatments have advanced, CD still leads to significant health issues due to disease progression and medication side effects. Exclusive enteral nutrition (EEN) is a recommended first-line treatment for pediatric CD, proving more effective than oral corticosteroids without side effects. However, EEN demands strict adherence, making it challenging for patients, particularly adults.

In 2019, Levine et al. found that a combination of a specific diet (CD exclusion diet, CDED) and partial enteral nutrition (PEN) was as effective as EEN in inducing remission in pediatric patients, with better tolerance and adherence. CDED focuses on whole foods and aims to minimize harmful dietary components affecting the gut.

In clinical practice, an adapted CDED (aCDED) has been used to provide more food choices, but it lacks validation in clinical trials. An aCDED that considers regional and seasonal food variations could enhance patient adherence and align with modern dietary preferences.

This study aims to compare the quality of life during a flare up of Crohn's disease treated with standard of care or an adapted Crohn's disease exclusion diet with partial enteral nutrition in adult patients.

DETAILED DESCRIPTION:
Crohn's disease (CD), a subgroup of inflammatory bowel disease (IBD), is increasing in incidence worldwide. Despite great advances in medical treatment, CD is associated with considerable morbidity related to progression of the chronic disease and the use of drugs that involve immunosuppression with an associated risk of serious infection as well as malignant and autoimmune sequelae.

Patients with CD often experience malnutrition due to factors like intestinal malabsorption, nutrient loss, restrictive diets, and increased energy expenditure during disease activity. Poor nutrition correlates with reduced treatment response and worse outcomes, emphasizing the significance of assessing and providing nutritional therapy in clinical practice. Additionally, CD is linked to elevated healthcare expenditures, diminished earning potential, comprised health-related metrics, and an overall reduction in quality of life.

In the management of CD, an emerging approach involves the exploration of nutritional interventions as an alternative to conventional therapy, which often entails medication regimes associated with potential side effects and risks.

Dietary therapy by means of exclusive enteral nutrition (EEN), consisting of a liquid formula diet excluding any other oral intake, has been shown to be superior to oral corticosteroids in induction of remission with no medical side effects, and is the recommended first-line treatment in pediatric patients with CD. However, EEN requires a firm commitment from the patients and their social environment to avoid any other oral food intake for 6 to 8 weeks, severely impeding therapy adherence and compliance.

In adult patients a Cochrane review showed a benefit of EEN. However, when the analysis was restricted to high-quality studies only, there was no difference between EEN and corticosteroids. Poor adherence to EEN by adults generally has reduced its utility as a key part of the therapeutic strategy.

An environmental hypothesis postulates that changes in dietary intake and industrialization of food contributes to the increasing incidence of IBD and CD. This is potentially due to alterations in the gut microbiome leading to impaired barrier function of the mucus layer and intestinal epithelium that is linked to processed foods. Therapies targeting the microbiome instead of primarily the immune system represent an attractive option that warrant further exploration. Diet appears to play a central role in the generation of inflammation by modulating the microbiome and intestinal barrier function. Plant-derived foods especially seem to shape the gut microbiome towards a more anti-inflammatory composition.

Different kinds of isocaloric partial enteral nutrition (PEN) with unrestricted exposure to food was not effective in reducing inflammation or inducing remission, suggesting that complete exclusion of food is key in the success of EEN.

EEN may therefore lead to remission both by the removal of specific dietary ingredients that trigger inflammation and by promoting a more anti-inflammatory microbiome. However, the absence of a more palatable and sustained dietary strategy that achieves the same results remains a main hurdle to the use of dietary therapy approaches in the wider IBD population.

In 2019, Levine et al showed that a restricted exclusion diet (Crohn's disease exclusion diet, in short CDED) combined with partial enteral nutrition (PEN) was similarly effective in remission induction to EEN in pediatric patients, while being better tolerated with a higher therapy adherence. CDED is a whole-food diet coupled with PEN, designed to reduce exposure to detrimental dietary components, hypothesized to negatively affect the microbiome, intestinal barrier function and intestinal immunity. It is characterized by a high amount of high-quality protein with reduced fat content and rich in complex carbohydrates whilst excluding certain components of the standard western diet. The combination with PEN, as a liquid formula, ensures a sufficient intake of calories with an extra supply of protein and vitamins [20]. Further clinical studies showed its efficacy in inducing clinical and endoscopic remission in adult patients with mild to moderate disease.

In clinical practice, the utilization of CDED is hampered because it is being restricted to very few food sources, with great differences in seasonal and regional availability. In addition, the protein intake in CDED relies heavily on animal protein, which does not meet contemporary diet styles and thus hampers adherence. The investigators propose a concept of an adapted CDED (aCDED) that respects regional and seasonal differences in food availability, thus improving patient adherence to the diet through better practicability, and also by meeting contemporary dietary requests. Through this the investigators expect to greatly increase the adherence and thus efficacy of this approach, particularly in adult patients. In comparison to standard CDED the aCDED is characterized by a higher amount of plant-derived protein with focus on minimally-processed items, a greater variety of fruits and vegetables and a more favorable omega 3 : 6 PUFA-ratio. This diet is complemented by Modulen, a liquid formula with optimal concentration of lipids, including a favorable omega 3 : 6 PUFA-ratio, and carbohydrates, vitamins and trace elements, which in concert have been shown to reduce intestinal inflammation in vitro and in vivo.

The combination of aCDED and Modulen aims to reduce the inflammation in the gut and promote gut mucosal healing by removing detrimental dietary components associated with inflammation and introducing beneficial food components that promote an anti-inflammatory gut microbiome. In addition, the diet aims to enhance the nutritional status of CD patients not only by mitigating inflammation but also by promoting improved nutrient absorption and utilization, ultimately supporting better nutritional outcomes, as suggested by several basic research efforts.

Patient's food choices and adherence to the diet will be evaluated using a questionnaire. Nutrition therapy in CD patients has been met by obstacles in previous studies, mainly due to poor therapy adherence. We tackle these issues by offering one-on-one nutrition counseling by trained personnel and will supply the patients with Modulen for the entire duration of the intervention phase. The nutritional status of the patients will be monitored during the study duration.

In summary, this approach provides a way for CD patients to manage their condition effectively, with a focus on nutrition and without the potential drawbacks of the standard medical treatment. It also emphasizes the importance of consistent dietary management as part of their overall strategy for dealing with the chronic condition.

As CD frequently afflicts young individuals, impeding their ability to work or pursue education, optimizing nutritional management as part of CD treatment can contribute to improved wellbeing and have further socioeconomic impact by means of cost savings in medical treatments as well as reduced days missing from work or university for IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥ 18 years at the time of signing the informed consent.
* Macroscopic small bowel involvement, or isolated large bowel disease confined to the right or transverse colon confirmed by endoscopy
* Patients with a Crohn's disease activity index (CDAI) of ≥ 150
* Patients will not be excluded if they have received 5ASA or an immunomodulator for > 8 weeks and the dose is stable, or if they start a thiopurine concurrently, as thiopurines are not considered sufficient to induce remission in active disease before 8 weeks as an isolated therapy
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures
* Able to adhere to the study visit schedule and other protocol requirements
* All subjects must agree to refrain from donating blood while on study drugs
* All subjects must agree not to share medication.
* Subject (male or female) is willing to use highly effective contraceptive methods during treatment and for 28 days (male or female) after the end of treatment

Exclusion Criteria:

* Patients with with minimal disease activity (CDAI <150) or severe disease (CDAI >450)
* Patients who have received corticosteroids of any kind in the previous 4 weeks
* Patients who have started an immunomodulator in the previous 8 weeks
* Any current biological or small molecule treatment
* Isolated large bowel disease iinvolving the recto-sigmoid or descending colon
* Patients with penetrating disease (abscess or fistula)
* Active perianal disease
* Fixed stricture or small bowel obstruction
* Normal fecal calprotectin
* Active extraintestinal disease (e.g. joint disease)
* Patients who have undergone an intestinal resection
* Sclerosing cholangitis
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
* Women during pregnancy and lactation Participation in other clinical trials or observation period of competing trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of Quality of Life | 12 weeks
  Measuring Quality of Life (QoL) using the IBD-Q-32-questionnaire (Inflammatory Bowel Disease Questionnaire with 32 items)
  * measuring the relative improvement compared to baseline
  * Minimum score: 32 points = bad QoL
  * Maximum score: 224 points = excellent QoL

SECONDARY OUTCOMES:
Remission (defined as CDAI≤150) | weeks 6, 12 and 24
  Using the CDAI (Crohn's Disease Activity Index) to measure activity in the past 7 days
  * score < 150 points = remission
  * score 150-219 points = mild disease activity
  * score 220-450 points = moderate to severe disease activity
  * score > 450 points = severe disease activity
Reduced fecal calprotectin | week 12 and 24
Patients' adherence to the diet assessed by cessation of therapy because of patients' refusal to continue and by a questionnaire | 12 weeks
Improvement of markers of malnutrition compared between the treatment arms | 12 weeks
Alterations in the microbiome in responders vs non-responders | 12 weeks
  - to assess changes in the oral and gut microbiome composition in responders vs non-responders oral (oral swab), fecal (stool kit) and tissue (endoscopy) and local microbiome (endoscopy) will be collected and genome sequencing will be performed
Alterations in the metabolome in responders vs non-responders | 12 weeks
  - to show alterations in the metabolome untargeted metabolomics from serum and fecal samples will be performed
Alterations in the intestinal immune profile in responders vs non-responders | 12 weeks
  - assessing the intestinal immune profile in responders vs non-responders through high dimensional immunoprofling (MACSIMA = mass cytometry by time-of-flight with single-cell in-drop massively parallel imaging) from tissue (endoscopy) provides a comprehensive analysis of the immune cell populations and their functional characteristics at the single-cell level. The simultaneous measure of multiple protein markers on individual immune cells allows a detailed examination of the immune system's composition and activity.
Link between genetic risk, microbiome, metabolome, intestinal immune profile and therapy outcome | 12 weeks
  * creating a link between results from extracting DNA from PBMC's from blood samples, microbiome composition, metabolome and therapy outcome as part of a personalised therapy approach
  * the assessment of the genetic risk will be performed by hotspot-analysis of the TLR5 gene
Measuring adverse events from steroid therapy | 12 weeks
  * Using the Streoid PRO Questionnaire (Patient-Reported Outcomes for Steroid Toxicity)
  * Measuring treatment-specific patientreported outcome measure for the impact of glucocorticoids from the patient perspective
  * higher score = more adverse events under steroid therapy
  * lower score = less adverse events under steroid therapy
Measuring mucosal inflammation | 12 weeks
  - using an endoscopic activity score (tba) and pathology findings

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Büringer, MD, Principal Investigator — Head of Department of Inflammatory Bowel Disease/Endoscopy
Locations (1):
- Universitätsklinik Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
All analyses will be performed in house in the university hospital of Tuebingen